CLINICAL TRIAL: NCT04930081
Title: The Effectiveness and Underlying Mechanisms of Parent Management Training and Mindful Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EA210088
Record Dates: First submitted 2021-06-10; First posted 2021-06-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-09

CONDITIONS: Parent Management Training; Mindfulness; Mindful Parenting Training
Keywords: Parent management training; Mindfulness; Parenting; Mindful parenting training; Parenting intervention; Parental support

STUDY DESIGN:
Intervention Model Description: A randomized-controlled design will be adopted. There will be two intervention groups, i.e. PMT and the MP programme, and one waitlist-control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants do not have knowledge of the interventions assigned to individual participants.
  The research assistant who supports in data collection do not know the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parent Management Training (Experimental): The well-researched Postivie Parenting Program (Triple P) is selected as the intervention program for the parent management training arm. It is an 8-week program that aims at equipping parents with effective parenting strategies.
  Interventions: Behavioral: Positive Parenting Program, Mindful Parenting
- Mindful Parenting Program (Experimental): The Mindful Parenting program, developed by Prof Susan Bogel is selected as the intervention program for the mindful parenting arm. It is an 8-week program that trains parents in mindfulness and support them to apply mindfulness in the parenting context.
  Interventions: Behavioral: Positive Parenting Program, Mindful Parenting
- Waitlist Control Group (No Intervention): The waitlist control group will not receive any service until two months after the intervention arms complete their training. Depending of the availability of the program instructor, either the Parent Management Training or the Mindful Parenting program will be offered to this group.

INTERVENTIONS:
Behavioral: Positive Parenting Program, Mindful Parenting — The Positive Parenting Program (Triple P) consists of 5 weekly group sessions (each lasting for 2 hours) plus three weekly individual telephone interview sessions (each lasting for around 20 minutes). Program materials is available in Chinese.
  The Mindful Parenting program consists of 8 weekly group sessions, each lasting for 2 hours. Programme materials have already been translated into Chinese by local partners of the programme developer.
  Arms: Mindful Parenting Program; Parent Management Training

SUMMARY:
Project Objective:

Parent management training (PMT), which focuses on teaching parents about effective discipline technique using a behavioral approach, has strong evidence base for promoting parent-child relationship, and reducing parental stress and children behavioural problem. Many PMTs, such as the Incredible Years and Triple P program, have been rated as well-established interventions for behavior problems in children.

In recent years, the application of mindfulness in the parenting context is emerging. Parental mindfulness was found to have positive effects on parent-child relationship quality and parenting stress. In particular, preliminary evidence of the eight-week mindfulness based intervention for parents, the Mindful Parenting (MP) program was found to reduce parental stress, and to decrease externalizing and internalizing problems in children.

The two lines of parenting intervention have different theoretical background but they yield similar positive effect in parents and children. The current study has the following objectives:

1. To explore the similarities and differences of PMT and MP in terms treatment outcome. Outcome measures include parenting knowledge, parent's mindful awareness, parents' emotional competence, positive and negative parenting practice, parental stress,parent-child relationship, and parents' mental health, including parental stress, parents' sense of competence, as well as child behavioural problem
2. To explore the underlying mechanisms for the effectiveness of PMT and MP, including their similarities and differences, and
3. To examine for whom are PMT and MP more effective.

Hypotheses

In terms of treatment outcome, it is hypothesized that:

H1a) When compared to the waitlist control group, both PMT and MP programmes are similarly effective in reducing negative parenting behaviours and behavioural problems in children, promoting positive parenting behaviours, and enhancing parent-child relationship and parents' mental health.

H1b) Looking into the different aspects of parenting behaviours, however, PMT has stronger effects than the MP programme on increasing proactive parenting and the use of positive reinforcement, and reducing lax control. By contrast, the MP programme has stronger effects than the PMT on enhancing warmth and supportiveness and reducing parental hostility.

In terms of mechanisms of change, it is hypothesized that:

H2a) The PMT and MP programmes both have positive effects on parents' mental health by way of improved parenting practices, and such effect is mediated by the reduction in child behavioural problems and improvement in parent-child relationship.

H2b) The PMT and MP programmes are different in how they bring about improved parenting practices. Parenting knowledge is the mediator between the PMT programme and improved parenting practices, whereas parent's emotional competence is the mediator between MP programme and improved parenting practices.

Lastly, in terms of the effectiveness for particular target participants, it is hypothesized that:

H3) PMT is less effective for parents with low emotional competence whereas the MP programme is more effective for parents with low emotional competence.

DETAILED DESCRIPTION:
Parental Influence on Child Development

It is not surprising that parents, who set the climate in the home environment, have large impact on the behavioural and emotional development in children. Numerous studies have shown that children of parents who are warm and responsive are more likely to experience optimal child development outcomes. On the contrary, timid, permissive and reactive parenting is found to be associated with emotional and behavioural difficulties in children.

Parent Management Training

Given the significant role that parents play, how to support parents become a matter of concern. Parent Management Trainings (PMT) have been demonstrated to be an effective form of parental support. Traditional PMTs are generally based on a behavioural approach, with a primary focus on educating parents on effective behavioural management strategies so as to induce changes in child behaviour.

Past research has proven that PMT is particularly effective for addressing emotional and behavioural difficulties in children. In a review of evidence-based treatment, PMT was found to gain the strongest empirical support and yield the largest effect size among all other treatment approaches for disruptive behaviours in children and adolescents. Programmes of this type include the Incredible Years (IY) Parent Programme, and Positive Parenting Programme (Triple P), which are both classified as 'Well-supported' programme in California Evidence-based Clearinghouse (https://www.cebc4cw.org/) and proven to be clinically effective and cost effective for training parents of children with significant behavioural problems. Outcome evaluation of PMT suggests that PMT yields the following positive results:

1. Increase in positive parenting behaviours, including more child-directed play, coaching and praise and reduced use of criticism and negative commands.
2. Increase in the use of effective limit-setting and replacing spanking and harsh discipline with proactive discipline techniques.
3. Increase in parental sense of competence and improve parent-child relationship.
4. Reduction in parental stress and child behavioural problems.

Mechanism of Parent Management Training

Although the effectiveness of PMT is well documented, the underlying mechanism of change for PMT is somewhat unclear. The effectiveness of PMT is likely accounted for by changes in parenting skills and behaviours, and associated with changes in parental self-efficacy, confidence, and attributions. Theoretically, it is assumed that parental behavioural change is itself a product of the knowledge of effective parenting practices acquired during PMT. For instance, knowledge of effective parenting strategies has been shown to be predictive of parenting competence, parent psychopathology, and child behavioural problems in a non-clinical sample. However, it could also be argued that while parents may understand what they "should" and what they "could" do, this knowledge may not necessarily translate into behaviour because of other factors, such as parental stress and parent's sense of competence. Overall, there is relatively little research examining the mechanism underlying the effectiveness of PMT and the role of parenting knowledge in these interventions. Further research is needed to examine the limitations and processes through which parenting knowledge may lead to the positive outcomes yielded by PMT.

Limitations of Parent Management Training

Despite the well-documented benefits of PMT programme, it was found that parents' capacity to regulate their own emotional arousal may influence the efficacy of the training. Others also argued that parents' ability in managing negative emotions plays a prominent role in parenting, but this is often not directly addressed in parent training programmes. Parent's own emotional competence, which broadly encompasses the ability to become aware of, recognize, accept, interpret, and respond constructively to one's own emotion, is central to the effective use of parenting skills because it affects the parent's capacity to respond to their child's behaviours in containing and sensitive ways, and reduces their hostile and coercive reactions. Parents with poor emotional competence, even after they have been equipped with effective parenting strategies, may have difficulty executing the strategies in the heat of the moment. Some researchers also posited that in times of high affective arousal, parents may have more difficulties in applying the newly acquired skills and therefore return to use the less skillful approach to manage their children. Moreover, anecdotal evidence of the author as a frontline service provider also confirms the above. Participants in PMT groups often reported that they were more confident in being parents upon programme completion because they had acquired effective parenting strategies. Nevertheless, some participants indicated that whether or not they could apply what they have learnt depends heavily on their ability to regulate their emotions. In other words, whether they could stay calm in times of parent-child conflict is a key factor.

Overall, there is a need to address parents' emotional processes in parental intervention and improving parental emotion regulation could be one avenue to help more parents.

Mindfulness and Parenting

Mindfulness is 'the awareness that emerges through paying attention on purpose, in the present moment, and non-judgmentally to the unfolding of experience moment by moment'. It can improve one's attention, promote tolerance to unpleasant sensations, feelings and thoughts; and can facilitate cognitive changes. It can also enhance the ability to cope with life challenges, through relaxation and facing difficulties with openness, and better management of caregiving duties. In the parenting context, high level of parental mindfulness is found to be associated with lower levels of parental stress and negative parenting behaviours (i.e. laxness, overreactivity, and verbosity) and increased adaptive parenting.

Given the numerous research which indicated that the practice of mindfulness could enhance resilience to emotional disturbances, and reduce emotional reactivity, mindfulness offers a promising direction for improving parental emotional competence.

Various researchers have proposed how mindfulness could be incorporated into the parenting context. For instance, it was suggested that parents can use mindfulness techniques to listen more openly to their children, develop emotional awareness, and better regulate their own emotions before reacting. Others also stated that in times of intense conflict, the practice of mindfulness could increase parents' parasympathetic tone so that they could be more focused and remain calm. The calmer and more mindful state of the parents could then facilitate parents to make wise choice in managing their children. Simply put, the practice of mindfulness may help transform reactive parenting to responsive parenting.

Recent research that investigates the effectiveness of mindfulnesss-based parenting programme yields positive results in general, supporting the utility of mindfulness in parenting. To date, mindfulness-based parenting programmes are reported to be effective in various populations, from parents of children with developmental delays, parents of children with special needs, to parents of early adolescents. Treatment effects include reducing negative mother-child interactions, decreasing mothers' emotional reactivity, and increasing parents' awareness of own emotions. In a local study, parents reported reduction in parental stress and depression, and improvement in emotion management after completion of a mindful parenting prorgamme. In general, teaching mindfulness practices to parents was effective in reducing child behavioural problems, enhancing parent-child relationship and enhances parents' well-being.

The Mindful Parenting (MP) Program

Literature reveals that the 'Mindful Parenting' (MP) programme, developed by Prof Susan Bögels in the Netherland, is one of the most extensively researched mindful parenting training to date. It is a new application of mindfulness which aims to improve parenting by improving the quality of parental attention, increasing awareness of parental stress, reducing parental reactivity, and decreasing the intergenerational transmission of dysfunctional parenting.

The MP programme is an eight-week mindfulness training for parents. It is an adaptation of the Mindfulness-Based Cognitive Therapy (MBCT) for depression, and the Mindfulness-Based Stress Reduction (MBSR) programme. The programme retains the basic structure and mindfulness practices of the MBCT and MBSR programs, but with a focus on the parenting context. Components specific to MP programme include automatic pilot parenting, parental self-compassion, and beginners mind parenting. Parents are also invited to apply mindfulness to interactions with their children, other family members, and the everyday tasks associated with parenting.

Research of the MP programme yields encouraging results. Parents who completed the programme reported an increase in mindful parenting, a reduction in negative parenting behaviours (including control, overreactivity, overprotection, and rejection), and an increase in positive parenting behaviours (including autonomy granting behaviour. Benefits to parental psychopathology and well-being include decreased stress and decreased internalizing and externalizing problems. In addition, the programme also brings positive impact to child's psychopathology, including decreased externalizing and internalizing problems.

Mechanism of the Mindful Parenting (MP) Programme

Given the encouraging preliminary evidence of the MP programme, how exactly does Mindful Parenting (MP) training work? What are the possible underlying mechanisms? There are six mechanisms of change through which the MP programme may improve parenting. They include:

1. Reducing parental stress and reactivity under stress.
2. Helping parents to embrace experiences with openness.
3. Improving parents' executive functioning in stressful and impulsive situations.
4. Recognizing and breaking cycle of intergenerational transmission of dysfunctional parenting schemas and habits.
5. Promoting attention that can increase care and compassion of self and the child.
6. Improving marital functioning and co-parenting.

Preliminary evidence was found to support that the MP works through 1) reducing parental stress and the assumed effect on parental reactivity and 2) improving marital functioning and co-parenting. In a more recent study, it was found that the programme made improvement in the area of parental stress, parenting, and co-parenting, but not on marital functioning. Putting together the above research results, the first pathway (i.e., reducing parental stress and the reactivity under stress) appeared to be the most strongly supported mechanism of change in the MP programme.

The well documented positive impact of mindfulness-based interventions on emotion regulation also supports this mechanism of change. With lowered emotion reactivity and improved functioning in stressful and emotionally charged situations, parents will have an increased capacity to tackle the parenting difficulties more skilfully, and thus reduce the use of negative parenting practice. Overall, it is probable that MP works through enhancing parental emotional competence, by reducing parent's reactivity and improving their functioning in stressful situations.

The Current Study

As described above, while there has been extensive research on the effectiveness and development of PMT, the MP programme is relatively less explored. The two lines of approaches are entirely different. For instance, while PMT primarily focuses on parent child interaction processes, the MP programme primarily focuses on changing parent's own emotional processes. Nevertheless, research evidence shows that the two lines of intervention yield similar treatment effects. In particular, they are both effective in improving parent's mental health (e.g., parental stress), reducing child behavioural problems, and improving parent-child relationship. Questions arise. How are the two programmes similar and different from each other in terms of treatment effects? What are the similarities and differences in their mechanisms of change? For whom are PMT and the MP programme more effective, or is there a difference?

To date, there are limited studies comparing the PMT and the MP programme. The current study sets out to address the above research gaps. In short, the current study intends to 1) explore the similarities and differences of PMT and the MP programme in terms of treatment outcomes, 2) explore the mechanisms underlying the effectiveness of PMT and the MP programme, and 3) examine for whom PMT and the MP programme are more effective. The hypotheses in the current study are listed below.

In terms of treatment outcome, it is hypothesized that:

H1a. When compared to the waitlist-control group, both PMT and MP programmes are similarly effective in reducing negative parenting behaviours and behavioural problems in children, promoting positive parenting behaviours, and enhancing parent-child relationship and parents' mental health.

H1b. Looking into the different aspects of parenting behaviours, however, PMT has stronger effects than the MP programme on increasing proactive parenting and the use of positive reinforcement, and reducing lax control. By contrast, the MP programme has stronger effects than the PMT on enhancing warmth and supportiveness and reducing parental hostility.

In terms of mechanisms of change, it is hypothesized that:

H2a. The PMT and MP programmes both have positive effects on parents' mental health by way of improved parenting practices, and such effect is mediated by the reduction in child behavioural problems and improvement in parent-child relationship.

H2b. The PMT and MP programmes are different in how they bring about improved parenting practices. Parenting knowledge is the mediator between the PMT programme and improved parenting practices, whereas parent's emotional competence is the mediator between MP programme and improved parenting practices.

Lastly, in terms of the effectiveness for particular target participants, it is hypothesized that:

H3. PMT is less effective for parents with low emotional competence whereas the MP programme is more effective for parents with low emotional competence.

ELIGIBILITY:
Inclusion Criteria:

* having children aged 6 to 12 years.

Exclusion Criteria:

* parents having a history of major mental illnesses and
* parents who have received 8 week parent management trainings or mindfulness courses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Parental Stress | Pre-intervention
  Parental Stress Scale (PSS) [Min. Value: 1; Max Value: 6 (with higher scores indicating higher levels of parental stress)]
Parental Stress | Post-intervention (Immediate)
  Parental Stress Scale (PSS) [Min. Value: 1; Max Value: 6 (with higher scores indicating higher levels of parental stress)]
Parenting Sense of Competence | Pre-intervention
  Parenting Sense of Competence Scale (PSOC) [Min. Value: 1; Max Value: 6 (with higher scores indicating higher parenting sense of competency)]
Parenting Sense of Competence | Post-intervention (Immediate)
  Parenting Sense of Competence Scale (PSOC) [Min. Value: 1; Max Value: 6 (with higher scores indicating higher parenting sense of competency)]
Parenting Sense of Competence | Delayed post-intervention (2 months follow-up)
  Parenting Sense of Competence Scale (PSOC) [Min. Value: 1; Max Value: 6 (with higher scores indicating higher parenting sense of competency)]
Parenting Behaviours | Pre-intervention
  Multidimensional Assessment of Parenting Scale (MAPS) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parenting behaviours in the particular subscale)]
Parenting Behaviours | Post-intervention (Immediate)
  Multidimensional Assessment of Parenting Scale (MAPS) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parenting behaviours in the particular subscale)]
Parenting Behaviours | Delayed post-intervention (2 months follow-up)
  Multidimensional Assessment of Parenting Scale (MAPS) [Min. Value: 1; Max Value: 5 (with higher score indicating higher frequency of the parenting behaviours in the particular subscale)]
Parent-Child Relationship | Pre-intervention
  Parent-Child Relationship Factor in the Parenting and Family Adjustment Scales (PAFAS) [Min. Value: 0; Max Value: 3 (with higher score indicating better parent child relationship)]
Parent-Child Relationship | Post-intervention (Immediate)
  Parent-Child Relationship Factor in the Parenting and Family Adjustment Scales (PAFAS) [Min. Value: 0; Max Value: 3 (with higher score indicating better parent child relationship)]
Parent-Child Relationship | Delayed post-intervention (2 months follow-up)
  Parent-Child Relationship Factor in the Parenting and Family Adjustment Scales (PAFAS) [Min. Value: 0; Max Value: 3 (with higher score indicating better parent child relationship)]
Child Behaviours | Pre-intervention
  Eyberg Child Behavior Inventory (ECBI) [Intensity Score: Min. Value: 1; Max Value: 7; Problem score: Min Value: 0; Max Value: 1 (with higher score indicating more child behavioral problem)]
Child Behaviours | Post-intervention (Immediate)
  Eyberg Child Behavior Inventory (ECBI) [Intensity Score: Min. Value: 1; Max Value: 7; Problem score: Min Value: 0; Max Value: 1 (with higher score indicating more child behavioral problem)]
Child Behaviours | Delayed post-intervention (2 months follow-up)
  Eyberg Child Behavior Inventory (ECBI) [Intensity Score: Min. Value: 1; Max Value: 7; Problem score: Min Value: 0; Max Value: 1 (with higher score indicating more child behavioral problem)]

SECONDARY OUTCOMES:
Parenting Knowledge | Pre-intervention
  Knowledge of Parenting Strategies Scale (KOPSS) (Brief Version) [Multiple Choice Questions, with four options in each question]
Parenting Knowledge | Post-intervention (Immediate)
  Knowledge of Parenting Strategies Scale (KOPSS) (Brief Version) [Multiple Choice Questions, with four options in each question]
Parenting Knowledge | Delayed post-intervention (2 months follow-up)
  Knowledge of Parenting Strategies Scale (KOPSS) (Brief Version) [Multiple Choice Questions, with four options in each question]
Parent's Emotional Competence | Pre-intervention
  Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating lower emotional competence)]
Parent's Emotional Competence | Post-intervention (Immediate)
  Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating lower emotional competence)]
Parent's Emotional Competence | Delayed post-intervention (2 months follow-up)
  Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) [Min. Value: 1; Max Value: 5 (with higher score indicating lower emotional competence)]
Mindful Parenting | Pre-intervention
  Interpersonal Mindfulness in Parenting (IM-P) [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of mindful parenting)]
Mindful Parenting | Post-intervention (Immediate)
  Interpersonal Mindfulness in Parenting (IM-P) [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of mindful parenting)]
Mindful Parenting | Delayed post-intervention (2 months follow-up)
  Interpersonal Mindfulness in Parenting (IM-P) [Min. Value: 1; Max Value: 5 (with higher score indicating higher level of mindful parenting)]

CONTACTS AND LOCATIONS:
Overall Officials: Hong Wang Denis Kwan, Master, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - H.K.T.A. Shun Yeung Primary School, Hong Kong
  - SKH Kei Fook Primary School, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided

REFERENCES:
- [Background] Beer, M., Ward, L., & Moar, K. (2013). The Relationship Between Mindful Parenting and Distress in Parents of Children with an Autism Spectrum Disorder. Mindfulness, 4(2), 102-112. Benn, R., Akiva, T., Arel, S., & Roeser, R. (2012). Mindfulness Training Effects for Parents and Educators of Children With Special Needs. Developmental Psychology, 48(5), 1476-1487. Bogels, S. (2013). MYmind mindfulness for children and adolescents with ADHD: therapist's manual. Amsterdam: University of Amsterdam. Bögels, S., Hellemans, J., Deursen, S., Römer, M., & Meulen, R. (2014). Mindful Parenting in Mental Health Care: Effects on Parental and Child Psychopathology, Parental Stress, Parenting, Coparenting, and Marital Functioning. Mindfulness, 5(5), 536-551. Bögels, S., & Restifo, K. (2014). Mindful parenting : A guide for mental health practitioners (Mindfulness in behavioral health). New York: Springer. Cheung, S. (2000). Psychometric properties of the Chinese version of the parental stress scale. Psychologia: An International Journal of Psychology in the Orient, 43, 253-253. Chorpita, B., Daleiden, E., Ebesutani, C., Young, J., Becker, K., Nakamura, B., . . . Starace, N. (2011). Evidence-Based Treatments for Children and Adolescents: An Updated Review of Indicators of Efficacy and Effectiveness. Clinical Psychology: Science and Practice, 18(2), 154-172. De Bruin, E. I., Zijlstra, B. J., Geurtzen, N., van Zundert, R. M., van de Weijer-Bergsma, E., Hartman, E. E., Nieuwesteeg, A. M., Duncan, L. G., & Bögels, S. M. (2014). Mindful parenting assessed further: Psychometric properties of the Dutch version of the Interpersonal Mindfulness in Parenting Scale (IM-P). Mindfulness, 5, 200-212. Duncan, L. G. (2007). Assessment of mindful parenting among families of early adolescents: development and validation of the Interpersonal Mindfulness in Parenting Scale (unpublished dissertation). Pennsylvania State University, University Park. Eyberg, S. M., & Ross, A. W. (1978). Assessment of child behavior problems: The validation of a new inventory. Journal of Clinical Child Psychology, 7(2), 113-116. Gibaud-Wallston, J., & Wandersman, L. P. (1978). Development and utility of the Parenting Sense of Competence Scale. Paper presented at the meeting of the American Psychological Association, Toronto, Canada. Kabat-Zinn, J. (2003). Mindfulness-based interventions in context: Past, present, and future. Clinical Psychology: Science and Practice, 10(2), 144-156. Kaufman, E. A., Xia, M., Fosco, G., Yaptangco, M., Skidmore, C. R., & Crowell, S. E. (2016). The Difficulties in Emotion Regulation Scale Short Form (DERS-SF): Validation and Replication in Adolescent and Adult Samples. Journal of Psychopathology and Behavioral Assessment, 38(3), 443-455. Kirkman, J. J. L., Dadds, M. R., & Hawes, D. J. (2018). Development and Validation of the Knowledge of Parenting Strategies Scale: Measuring Effective Parenting Strategies. Journal of Child and Family Studies, 27(10), 3200-3217. Leung, C. M., Chan, S. C. M., Pang, R. C. Y., & Cheng, W. K. C. (2003). Validation of the Chinese version of the Eyberg child behaviour inventory for use in Hong Kong. Education and Manpower Bureau. Leung, C., & Tsang, S. K. M. (2010). The Chinese Parental Stress Scale: Psychometric Evidence Using Rasch Modeling on Clinical and Nonclinical Samples. Journal of Personality Assessment, 92(1), 26-34. Ngai, Fei-Wan, Chan, Wai-Chi Sally, & Holroyd, Eleanor. (2007). Translation and Validation of a Chinese Version of the Parenting Sense of Competence Scale in Chinese Mothers. Nursing Research (New York), 56(5), 348-354. Parent, J., & Forehand, R. (2017). The Multidimensional Assessment of Parenting Scale (MAPS): Development and Psychometric Properties. Journal of Child and Family Studies, 26(8), 2136-2151. Rochelle, Tina L, & Cheng, H T. (2016). Parenting Practices and Child Behaviour Problems in Hong Kong: Knowledge of Effective Parenting Strategies, Parenting Stress, and Child-Rearing Ideologies. Child Indicators Research, 9(1), 155-171. Sanders, M. R., Morawska, A., Haslam, D., Filus, A., & Fletcher, R. (2014). Parenting and Family Adjustment Scales (PAFAS): Validation of a brief parent-report measure for use in assessment of parenting skills and family relationships. Child Psychiatry & Human Development, 45, 255-272. Segal, Z. V., Williams, J. M. G., & Teasdale, J. D. (2002). Mindfulness-based cognitive therapy for depression: A new approach to preventing relapse. New York: Guilford. Siegel, D. J., & Hartzell, M. (2004). Parenting from the inside out: How a deeper self understanding can help you raise children who thrive. New York: Penguin. Singh, N. N., Lancioni, G. E., Winton, A. S. W., Singh, J., Curtis, W. J., Wahler, R. G., & Mcaleavey, K. M. (2007). Mindful Parenting Decreases Aggression and Increases Social Behavior in Children With Developmental Disabilities. Behavior Modification, 31(6), 749-771.